CLINICAL TRIAL: NCT00099619
Title: Efficacy of Exenatide Compared With Insulin Glargine in Patients With Type 2 Diabetes Using Metformin or Sulfonylurea for Whom Insulin is the Next Appropriate Therapy
Brief Title: Comparing Exenatide and Insulin Glargine in Type 2 Diabetes Patients for Whom Insulin is the Next Appropriate Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWAO
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; exendin-4; diabetes; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exenatide/insulin glargine (Experimental): Arm that first receives exenatide, then crosses over to insulin glargine
  Interventions: Drug: exenatide/insulin glargine
- Insulin glargine/exenatide (Experimental): Arm that first receives insulin glargine, then crosses over to exenatide
  Interventions: Drug: insulin glargine/exenatide

INTERVENTIONS:
Drug: exenatide/insulin glargine — Subcutaneously injected exenaide 10 mcg twice daily for 16 weeks; then insulin glargine subcutaneously injected once daily for 16 weeks given in a dose that varies for individuals to achieve target glucose levels
  Other Names: Byetta; AC2003; syntheitc exenden-4
  Arms: exenatide/insulin glargine
Drug: insulin glargine/exenatide — Subcutaneously injected insulin glargine subcutaneously injected once daily for 16 weeks given in a dose that varies for individuals to achieve target glucose levels; then exenaide 10 mcg twice daily for 16 weeks
  Other Names: Byetta; AC2993; synthetic exenden-4
  Arms: Insulin glargine/exenatide

SUMMARY:
This is a study with two treatment sequences and two treatment periods that will assess the safety and efficacy of exenatide treatment in patients with type 2 diabetes who have inadequate glycemic control using metformin or sulfonylurea and for whom insulin is the next appropriate step in diabetes treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Treated with a stable dose of metformin or sulfonylurea for at least 3 months prior to screening.
* HbA1c between 7.1% and 11.0%, inclusive.
* Insulin therapy should be the next appropriate step of diabetes treatment.
* Body Mass Index (BMI) >25 kg/m2 and <40 kg/m2.

Main Exclusion Criteria:

* Patient previously in a study involving exenatide or glucagon-like peptide-1 analogs.
* Treated with insulin, thiazolidinediones, alpha-glucosidase inhibitors, or meglitinides within 3 months prior to screening.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2004-09; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated hemoglobin) from the baseline of the first period (16-weeks of exenatide or insulin) to the end of each 16-week period. | Baseline, Week 16, Week 32
  Change in HbA1c from Baseline to the end of each 16-week period. There is one 16-week period of exenatide treatment and one 16-week period of insulin glargine.

SECONDARY OUTCOMES:
Change in patient-reported outcomes from Baseline to the end of each 16-week period | Baseline, Week 16, Week 32
  Change in patient-based outcomes (Hypoglycemic Fear Survey, patient-preference questionnaires [Treatment Evaluation and Treatment Preference questionnaires), Diabetes Symptom Checklist-Revised, Diabetes Treatment Flexibility Scale, Psychological General Well-Being Index, and the EuroQol (EQ-5D) instrument] from Baseline to the end of each 16-week exenatide or insulin glargine period

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (26):
- Australia (5):
  - Research Site, Westmead, New South Wales
  - Research Site, Daw Park, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, East Ringwood, Victoria
- Greece (3):
  - Research Site, Athens
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Pécs
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- Italy (6):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Perugia
  - Research Site, Rome
- Mexico (4):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Monterrey, N.l.
  - Research Site, Mexico City
- Poland (3):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Lublin

REFERENCES:
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356